CLINICAL TRIAL: NCT06304779
Title: The Effect of Continuous Intravenous Infusion of Lidocaine on Postoperative Pulmonary Complications and Prognosis in Emergency Surgical Patients With Intra-abdominal Infection
Brief Title: The Effect of Continuous Intravenous Infusion of Lidocaine on PPCs and Prognosis in Emergency Surgical Patients With IAI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V3.0.2023.11.29
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pulmonary Complications; Intra-abdominal Infection
Keywords: intra-abdominal infection; lidocaine; postoperative pulmonary complications
MeSH Terms: conditions — Intraabdominal Infections | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Lidocaine group: Patients receive a loading dose of 1.5 mg/kg 2% lidocaine at anesthesia induction, followed by continuous intravenous infusion at 1.5 mg/kg/h until 24 hours postoperatively Control group: Patients receive an equivalent volume of normal saline at anesthesia induction and throughout the perioperative period until 24 hours postoperatively.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Patients receive an equivalent volume of normal saline at anesthesia induction and throughout the perioperative period until 24 hours postoperatively.
  Interventions: Drug: Placebo
- Lidocaine group (Experimental): Patients receive a loading dose of 1.5 mg/kg 2% lidocaine at anesthesia induction, followed by continuous intravenous infusion at 1.5 mg/kg/h until 24 hours postoperatively.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine group receive a loading dose of 1.5 mg/kg 2% lidocaine at anesthesia induction, followed by continuous intravenous infusion at 1.5 mg/kg/h until 24 hours postoperatively and Control group receive an equivalent volume of normal saline at anesthesia induction and throughout the perioperative period until 24 hours postoperatively.
  Both groups will receive the same anesthesia and postoperative analgesia protocols, lung-protective ventilation strategy, and fluid, transfusion, and warming strategies. The only difference is the intervention during surgery, with the lidocaine group receiving continuous intravenous lidocaine.
  Arms: Lidocaine group
Drug: Placebo — atients receive an equivalent volume of normal saline at anesthesia induction and throughout the perioperative period until 24 hours postoperatively.
  Arms: Control group

SUMMARY:
The main purpose of this study is to evaluate the impact of continuous 24-hour intravenous infusion of lidocaine on the incidence of PPCs in patients undergoing emergency laparotomy for intra-abdominal infection (IAI).The secondary objectives of this study are to assess the impact of continuous 24-hour intravenous lidocaine infusion on the proportion of patients requiring mechanical ventilation, protection of important organ function during the perioperative period, length of hospital stay, and outcomes within 30 days postoperatively.

DETAILED DESCRIPTION:
PPCs are defined as the occurrence within 2 days postoperatively of atelectasis unplanned ventilation, acute respiratory distress syndrome (ARDS), and postoperative pneumonia syndrome Unplanned ventilation postoperatively: Defined as the use of non-invasive mechanical ventilation, invasive mechanical ventilation, or extracorporeal membrane oxygenation (ECMO) after the first extubation postoperatively or if extubation cannot be performed as planned.

Acute Respiratory Distress Syndrome (ARDS): Defined as acute diffuse inflammatory lung injury leading to increased pulmonary vascular permeability, increased lung weight, loss of aerated lung tissue, hypoxemia, and bilateral opacities on imaging (using the Berlin Consensus definition).

Postoperative pneumonia: Defined according to the diagnostic criteria in the "Chinese Adult Hospital-Acquired Pneumonia and Ventilator-Associated Pneumonia Diagnosis and Treatment Guidelines" (2018 version): new or progressive infiltrates, consolidation, or ground-glass opacities on chest X-ray or CT, along with two or more of the following clinical symptoms: ① fever (> 38.0°C), ② purulent respiratory secretions, ③ peripheral blood leukocyte count > 10×10^9/L or < 4×10^9/L.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, any gender.
* Patients suspected of digestive tract perforation or obstruction based on physical examination, confirmed by imaging, requiring emergency surgical treatment.
* The anesthesia method is general anesthesia
* I or the patient's family have carefully read and signed the informed consent form
* Serum procalcitonin (PCT) at inflammatory levels or leukocytosis (>12×109/L) or leukopenia (<4×109/L) or >10% naive leukocytes

Exclusion Criteria:

* Have a history of local anesthesia drug allergy
* Pregnant patients
* Patients receiving renal replacement therapy
* Patients with arrhythmias or heart failure (second or third-degree atrioventricular block or left ventricular ejection fraction [LVEF]
* Preoperative platelet count<80 × 109/L
* Patients who require secondary surgery for postoperative anastomotic fistula
* Patients who have participated in other clinical studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The impact of continuous 24-hour intravenous lidocaine on the incidence of PPCs in patients undergoing emergency laparotomy for IAI. | within 2 days after surgery
  PPCs are defined as a syndrome encompassing atelectasis, unplanned mechanical ventilation, acute respiratory distress syndrome (ARDS), and postoperative pneumonia occurring within 2 days after surgery.

SECONDARY OUTCOMES:
the impact of continuous 24-hour intravenous lidocaine infusion on the proportion of patients requiring mechanical ventilation, protection of important organ function during the perioperative period | within 30 days postoperatively
  The protection of important organ function during the perioperative period is defined as the difference in Sequential Organ Failure Assessment (SOFA) scores between the highest preoperative and postoperative 2-day scores (Delta-SOFA), following the "Sepsis 3.0 International Consensus on Sepsis and Septic Shock."

OTHER OUTCOMES:
To observe the impact of continuous perioperative lidocaine infusion on the levels of neutrophil extracellular traps (NETs) postoperatively | before anesthesia, 24 hours postoperatively, and 7 days postoperatively
  Twenty patients from each group will be selected for blood collection before anesthesia, 24 hours postoperatively, and 7 days postoperatively, to explore the potential mechanisms influencing peripheral blood NETs levels

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital,Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No